CLINICAL TRIAL: NCT04004169
Title: Closed-Loop Deep Brain Stimulation for Treatment-Resistant Depression
Brief Title: Closed-Loop Deep Brain Stimulation for Major Depression
Acronym: PReSiDio
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Andrew Krystal (Other)
Responsible Party: Sponsor-Investigator, Andrew Krystal, Professor of Psychiatry and Behavioral Sciences, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 17-23724
Record Dates: First submitted 2019-06-26; First posted 2019-07-01 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Depression; Treatment-resistance; Deep brain stimulation; Closed-loop; Biomarker; Responsive neurostimulation; Brain surgery
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Arm 1: Intervention (stimulation ON) (Experimental): This is a crossover trial. Each patient will receive 6 wks of stimulation ON (arm 1), stimulation OFF (arm 2), and Stimulation ON Active Control (sham biomarker) (arm 3) in random order. After 6 months of intervening therapy, this 3-period crossover study will be repeated.
  Interventions: Device: Stimulation-ON
- Arm 2: Sham Control (stimulation OFF) (Sham Comparator): This is a crossover trial. Each patient will receive 6 wks of stimulation ON (arm 1), stimulation OFF (arm 2), and Stimulation ON Active Control (sham biomarker) (arm 3) in random order. After 6 months of intervening therapy, this 3-period crossover study will be repeated.
  Interventions: Device: Stimulation-OFF
- Arm 3: Active Control (stimulation ON triggered by sham biomarker) (Active Comparator): This is a crossover trial. Each patient will receive 6 wks of stimulation ON (arm 1), stimulation OFF (arm 2), and stimulation ON Active Control (sham biomarker) (arm 3) in random order. After 6 months of intervening therapy, this 3-period crossover study will be repeated.
  Interventions: Device: Stimulation-ON Active Control

INTERVENTIONS:
Device: Stimulation-ON — Active neurostimulation from the NeuroPace RNS® System triggered by a biomarker
  Arms: Arm 1: Intervention (stimulation ON)
Device: Stimulation-OFF — No neurostimulation from the NeuroPace RNS® System
  Arms: Arm 2: Sham Control (stimulation OFF)
Device: Stimulation-ON Active Control — Active neurostimulation from the NeuroPace RNS® System triggered by a sham biomarker
  Arms: Arm 3: Active Control (stimulation ON triggered by sham biomarker)

SUMMARY:
Neurons are specialized types of cells that are responsible for carrying out the functions of the brain. Neurons communicate with electrical signals. In diseases such as major depression this electrical communication can go awry. One way to change brain function is using electrical stimulation to help alter the communication between groups of neurons in the brain.

The purpose of this study is to test a personalized approach to brain stimulation as an intervention for depression. The study researchers will use a surgically implanted device to measure each individual's brain activity related to his/her depression. The researchers will then use small electrical impulses to alter that brain activity and measure whether these changes help reduce depression symptoms. This study is intended for patients with major depression whose symptoms have not been adequately treated with currently available therapies.

The device used in this study is called the NeuroPace Responsive Neurostimulation (RNS) System. It is currently FDA approved to treat patients with epilepsy. The study will test whether personalized responsive neurostimulation can safely and effectively treat depression.

DETAILED DESCRIPTION:
This is a single-center 3-stage feasibility study of personalized closed-loop stimulation for treatment resistant Major Depressive Disorder. Depending on participant's results at each stage, he/she might not be eligible to proceed to all 3 stages.

Stage 1 of the study will involve surgically implanting small, thin electrodes in brain regions that regulate depression in order to identify personalized treatment sites. The researchers will test stimulation in the different brain regions and their effect on depression symptoms. The electrodes will be surgically removed at the end of Stage 1.

Stage 2 will involve a second brain surgery to implant the NeuroPace RNS® System. Researchers will use information from Stage 1 to decide where to implant the electrodes of the RNS System. Over the next ~4-12 months, participants will have regular study visits in the clinic where the researchers will determine a personalized brain activity pattern that correlates with depression symptoms and can be paired with stimulation to improve depression symptoms.

Stage 3 will be 12 months long and will involve turning ON and OFF the intervention to test its effectiveness. Over the course of a year, the participant will have two 6-week periods with no stimulation and will receive the intervention for the remainder of the time.

At the end of this stage the participant can choose to continue with long-term follow-up or have the RNS System surgically removed.

ELIGIBILITY:
Inclusion Criteria:

* Age 22-70
* Meet the Diagnostic and Statistical Manual of Mental Disorders (DSM-V) diagnostic criteria for Major Depressive Disorder (MDD) without psychosis based on a Structured Clinical Interview for DSM-V (SCID) with current episode ≥ 2 years that is treatment- resistant (4 adequate trials (including ECT), 3 classes of medications, one augmentation strategy, psychotherapy) as measured by the antidepressant treatment history form (ATHF).
* Failed electroconvulsive therapy (ECT) due to inability to achieve sustained response (2 failed attempts to discontinue ECT treatment) or discontinued due to intolerable side effects.
* Has MADRS score of > 26 at both baseline and screening visit
* The presence of variability on repeated administrations of MDD rating scales (minimum of 2-point variation on the HAMD-6 administered 3 times a day for 3 days), which is required for the identification of a neural biomarker.
* If patient is on a regimen of psychotropic medication, no changes in this regimen should be made during the 4 weeks prior to entry into and the duration of the study.
* Willing and able to undergo invasive brain recording/stimulation study
* Willing and able to attend multiple research visits and perform at-home research protocol
* Willing and able to provide informed consent
* Ability to speak and read English

Exclusion Criteria:

* Meets DSM-V criteria for a psychotic disorder, eating disorder, panic disorder, posttraumatic stress disorder, bipolar disorder, obsessive compulsive disorder, tic disorder, or another comorbid psychiatric disorder other than MDD or generalized anxiety disorder based on a SCID
* Generalized anxiety disorder is the primary DSM-V disorder during the current MDD episode
* Active suicidal ideation with intent and plan as defined by a score of 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS)
* History of suicide attempt requiring hospitalization in previous 2 years.
* Meets criteria for alcohol or substance abuse or dependence (other than caffeine) in previous 6 months, determined by the SCID
* Has a personality disorder based on the investigator's assessment that the investigator believes will adversely impact subject compliance or safety
* Fibromyalgia or chronic fatigue syndrome
* Current condition requiring chronic narcotic use
* History of traumatic brain injury, another neurological disorder, or developmental delay
* History of seizures
* MRI (done within one year of the first visit) with significant abnormalities
* Previous ablative intracranial surgery or previously implanted deep brain stimulation system or any previously implanted device treatment involving brain stimulation
* Implantable hardware not compatible with MRI or with the study
* Major medical co-morbidities increasing the risk of surgery including severe diabetes, major organ system failure, history of hemorrhagic stroke, need for chronic anticoagulation other than aspirin, active infection, intracranial space occupying lesion, increased intracranial pressure, cardiovascular accident within the last month, aneurysm/abnormality, retinal detachment, unstable cardiovascular disease (recent myocardial infarction, severe ischemia, severe or uncontrolled hypertension), immunocompromised state, or malignancy with < 5 years life expectancy
* Inability to stop Coumadin or platelet anti-aggregation therapy for surgery and after surgery. - Patients taking these medications will need to discuss the need/risk of continuing these medications with their physicians and the PI or study personnel may contact the treating physician(s) to discuss the risks of anticoagulation/antiaggregation therapy discontinuation
* Coagulopathy. Patients will be excluded unless assessed and cleared by hematology
* Allergies or known hypersensitivity to materials in the NeuroPace RNS® System (i.e. titanium, polyurethane, silicone, polyetherimide, stainless steel)
* Subject lives alone without possibility of caregiver support post-hospital stay
* Inability to comply with study follow-up visits
* Women who are pregnant, plan to become pregnant, or breast feeding
* Inability to speak and/or read English
* Inability to give consent
* Significant cognitive impairment or dementia (MoCA < 25)
* Likely to require ECT during the course of the study

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2019-07-18 (Actual); Primary Completion 2030-06-28 (Estimated); Study Completion 2035-06-28 (Estimated)

PRIMARY OUTCOMES:
change in MADRS score | administered at baseline and every 2 weeks for the first 18 weeks of stage 3
  Effect size of active compared to sham stimulation (mean difference in Montgomery Asberg Depression Rating Scale (MADRS) score before and after the sham and treatment periods). Higher MADRS score indicates more severe depression; the overall score ranges from 0 to 60.

SECONDARY OUTCOMES:
change in Montgomery Asberg Depression Rating Scale (MADRS) score after 1 year | administered at Weeks 30 and every 2 weeks for the last 18 weeks of Stage 3
  Effect size of active compared to sham stimulation (mean difference in Montgomery Asberg Depression Rating Scale (MADRS) score before and after the sham and treatment periods at the end of Stage 3. Higher MADRS score indicates more severe depression; the overall score ranges from 0 to 60.
difference in Hamilton Depression Rating Scale (HAMD-17) score | administered at baseline and every 2 weeks for the first 18 weeks of stage 3
  Mean difference in Hamilton Depression Rating Scale (HAMD-17) score across the two 6-week cross-over periods. The score for Hamilton Depression Rating Scale ranges from 0-50, with a higher score indicating more severe depression.
difference in Hamilton Depression Rating Scale (HAMD-17) score after 1 year | administered at Weeks 30 and every 2 weeks for the last 18 weeks of Stage 3
  Mean difference in Hamilton Depression Rating Scale (HAMD-17) score across the two 6-week cross-over periods at 1 year. The score for Hamilton Depression Rating Scale ranges from 0-50, with a higher score indicating more severe depression.
difference in the Inventory of Depressive Symptomatology Self-Report (IDS-SR) score | administered at baseline and every 2 weeks for the first 18 weeks of stage 3
  Mean difference in Inventory of Depressive Symptomatology Self-Report (IDS-SR) score across the two 6-week cross-over periods. The scores range from 0 to 27, with higher scores indicating more depressive symptoms.
difference in Inventory of Depressive Symptomatology Self-Report (IDS-SR) score after 1 year | administered at Weeks 30 and every 2 weeks for the last 18 weeks of Stage 3
  Mean difference in Inventory of Depressive Symptomatology Self-Report (IDS-SR) score across the two 6-week cross-over periods at the of Stage 3. The scores range from 0 to 27, with higher scores indicating more depressive symptoms.

OTHER OUTCOMES:
Stimulation site identification | Final study visit of Stage 1 (roughly 3-6 months after initial enrollment)
  Over 50% of patients move from Stage 1 to Stage 2 (stimulation site that acutely improved mood identified)
Biomarker identification in Stage 1 | Final study visit of Stage 1 (roughly 3-6 months after initial enrollment)
  The number of patients in whom we can identify a neural biomarker that accounts for a significant amount of variance in depression symptom severity
Number of patients who had viable biomarker(s) identified in Stage 2 | Final study visit of Stage 2 (up to 1 year duration)
  The number of patients in whom we can identify a neural biomarker utilizing the RNS system that accounts for a significant amount of variance in depression symptom severity
The number of patients in whom we can identify a neural biomarker utilizing the RNS system that accounts for a significant amount of variance in depression symptom severity | Assessed at the final study visit of Stage 3 (1 year duration)
  The number of patients in whom we can find a personalized biomarker of depression in terms of accounting for significant variance in depression
The number and type of serious adverse events for patients that occur in closed-loop deep brain stimulation with the device | Safety will be monitored continuously throughout the ~2 years of trial enrollment
  The number and type of serious adverse events that occur in comparison to comparable open-loop deep brain stimulation trials
Relationship of biomarkers identified in Stage 2 and Stage 1 | Assessed at the end of Stage 2 (up to 1.5 year duration)
  The number of subjects for whom the biomarker identified with Stage 1 data is able to be replicated in Stage 2 in terms of a measure obtained from the same recording site and in a comparable frequency range accounting for a significant amount of variance in depression severity.
Achievement of Long-Term Symptom Control | Assessed at end of Stage 3 (up to 1 year duration)
  Number of subjects who achieve long-term symptom control with treatment in terms of being in remission at the end of the 3 months of active therapy between the two randomized trials in Stage 3.
Non-inferiority of closed loop vs open-loop intermittent stimulation therapy and sham stimulation | administered at baseline and every 2 weeks for the first 18 weeks of stage 3
  Number of subjects for whom active closed-loop therapy is associated with equal or lower MADRS scores compared with: 1) active intermittent stimulation driven by a sham biomarker control and 2) sham stimulation control.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Krystal, MD, MS, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No